CLINICAL TRIAL: NCT01664988
Title: Effect of Muscular Relaxation and Breathing Technique on Blood Pressure in Pregnancy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, mahboobeh aalami, researcher, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: muscular relaxation
Record Dates: First submitted 2012-07-24; First posted 2012-08-15 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Blood Pressure in Pregnancy

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- muscular relaxation (Experimental): muscular relaxation was done using Jacobson by contracting and relaxing selected groups of muscles until total relaxation
  Interventions: Behavioral: muscular relaxation
- breath control (Experimental): include deep diaphragmatic breathing and decrease breath rate to 6-10/min
  Interventions: Behavioral: breath control
- control (Other): received routine care of clinic or health center and control their blood pressure weekly and use drugs if necessary
  Interventions: Other: control (routine care)

INTERVENTIONS:
Behavioral: muscular relaxation — muscular relaxation was done using Jacobson by contracting and relaxing selected groups of muscles until total relaxation
  Other Names: one
  Arms: muscular relaxation
Behavioral: breath control — breathing control techniques include deep diaphragmatic breathing and decrease breath rate to 6-10/min
  Other Names: two
  Arms: breath control
Other: control (routine care) — received routine care of clinic or health center and use drugs if necessary
  Other Names: 3
  Arms: control

SUMMARY:
Gestational hypertension is the main cause of maternal and fetal mortality, however, it has no definite effective treatment. nowadays, the stress management approaches are use for essential hypertension. So, this study aimed is study the effect of progressive muscular relaxation and breathing control technique on blood pressure during pregnancy.

this 3-groups clinical trial has been done in Mashhad Health Centers and Governmental hospitals. 60 pregnant women with systolic blood pressure less than 135 mm Hg or diastolic blood pressure more than 85 mm Hg who met inclusion criteria were assigned into three groups of progressive muscular relaxation, breathing control and control. In tow experiment groups, exercises were controlled by one day personally and the rest by CD, BP before and after interventions was controlled for 4 weeks. In control group blood pressure was measured before and after 15 minutes with no intervention.

ELIGIBILITY:
Inclusion Criteria:

* systolic blood pressure ≥ 135mmHg or
* diastolic blood pressure ≥ 85mmHg
* absence of severe preeclampsia condition
* eclampsia
* absence chronic hypertension
* gestational age 20-36w
* single pregnancy
* have not contraction or bleeding
* absence of underlying disease and mental disorders
* absence of polihydramnios
* hydatiform mole and placenta previa
* not addicted to drugs, alcohol, mood-altering medicine and cigarette
* not to use similar relaxation methods and breathing techniques during pregnancy
* reading and writing literacy
* have contact number

Exclusion Criteria:

* using antihypertensive drugs(for experimental groups)
* CBR
* bleeding
* contraction or watering during study
* deteriorating of preeclampsia to severe form
* hospitalization
* start medical treatment for experiment groups
* changing mind for continuing with study
* to be absent in one session of personal instruction for experiment groups do not exercises more than 3 sessions of relaxation and breathing control at home
* delivery during 4- week interventions and presence of symptoms such as confusion, fatigue, feeling of suffocation, pain, blurred vision during doing exercises

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
effect of muscular relaxation | up to1 month
  effect of muscular relaxation by check of the blood pressure after muscular relaxation was controlled
decrease blood pressure | up to 1 month

SECONDARY OUTCOMES:
time of decreasing blood pressure | up to 1 month